CLINICAL TRIAL: NCT04741815
Title: The Effect of Different Warming Methods Applied to Patients for Prevention of Hypothermia on Pain, Comfort and Some Parameters in Laparoscopic Cholecystectomy Surgery
Brief Title: Effects of Different Warming Methods in Laparoscopic Cholecystectomy Surgery
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Bozok University (Other)
Collaborators: Ataturk University (Other)
Responsible Party: Principal Investigator, Aybike Bahçeli, Research Asistant, Bozok University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: 2018-3/16
Record Dates: First submitted 2021-01-27; First posted 2021-02-05 (Actual); Last update posted 2022-03-02 (Actual); Status verified 2022-02

CONDITIONS: Inadvertent Perioperative Hypothermia
Keywords: Inadvertent Perioperative Hypothermia; laparoscopic cholecystectomy; nurse; pain; physiological parameters; shivering; thermal comfort
MeSH Terms: conditions — Pain

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Forced Air Warming Group (Experimental): There is no intervention in patients before the operation. When he comes out of the operation and comes to the post-anesthesia care unit (PACU), he is warmed by forced air. When the body temperature of the patients reaches 36 ° C, they are transferred to the clinic with a cover and blanket.
  Interventions: Device: Forced Air Warming
- Peripheral Carbon Fiber Warming Group (Experimental): Gloves and socks developed by the researcher are applied half an hour before the operation. These materials, called environmental warming, have three layers. The first layer in contact with the patient is a thermal inner sheath made of 90% Polyester and 10% Polyamide and is used to maintain body temperature. The second layer consists of carbon fiber warmer and foil. The end of the carbon fiber warmer is USB connected. When the connection is plugged in, the warmer works. The third layer is again made of thermal fabric. A rubber bandage is made to separate the last layer from the external environment and to maintain the patient's body temperature. The USB connection is removed while patients are sent for surgery. After the operation, rewarming is started in the post-anesthesia care unit. When the patient's body temperature reaches 36 ° C, he is transferred to the clinic with a cover and blanket.
  Interventions: Device: Peripheral Carbon Fiber Warming
- Control Group (No Intervention): A routine hospital procedure is applied. The patient is not warmed before going to surgery. A cover and blanket are used passively after being taken to the PACU from the operation.

INTERVENTIONS:
Device: Forced Air Warming — It consists of the WarmAir® unit and FilteredFlo® blankets. FilteredFlo® blankets are a cover designed to cover the entire body and extremities with air channels that provide the appropriate distribution of patient warm. The WarmAir® warming device connected to the shroud via a pipe; it has three temperature settings, 32.2 C, 37.8 C, and 43.3 C.
  Arms: Forced Air Warming Group
Device: Peripheral Carbon Fiber Warming — It was developed by the researcher. Designed as gloves and socks, these warming materials have three layers. The first layer in contact with the patient and the third layer in contact with the external environment is a thermal material to maintain body temperature. The second floor consists of a USB-connected carbon fiber warmer and foil.
  Arms: Peripheral Carbon Fiber Warming Group

SUMMARY:
Cold gases given during laparoscopic cholecystectomy are the most important cause of hypothermia. However, even surgery alone is an 80% important cause of hypothermia. Inadvertent perioperative hypothermia is a common complication of the surgical process that can cause serious complications. In most of the patients, tremors, increase in pain, deterioration in comfort and changes in some physiological parameters can be seen. Despite this, there are not enough warming devices that nurses can use practically and are easy to use, affordable and comfortable for the patient. In the literature, it is stated in the evidence-based guidelines for determining the hypothermia risks of patients and taking early precautions.

DETAILED DESCRIPTION:
The parallel group randomized controlled three group study blinded by the evaluator aims to investigate the effectiveness of different warming methods in laparoscopic cholecystectomy patients. This study general surgery at Yozgat Bozok University Hospital in Turkey are performed in clinics. All patients are male and female patients who have undergone surgery and met the inclusion criteria.

ELIGIBILITY:
Inclusion Criteria:

* Patients are qualified to answer research questions,
* BMI is between 18.5 kg / m2 and 30 kg / m2,
* Not using therapeutic hypothermia in the surgery,
* Not being treated with chronic opioids,
* Operation time is between 60 minutes and 6 hours,
* Having received general anesthesia during the operation,
* Reception of patients with ASA classification I or II,
* Absence of anemia, coagulation problem and peripheral circulatory disease or metabolic disease.

Exclusion Criteria:

* Intraoperative and postoperative have complications (bleeding, arrest, nausea, vomiting, etc.),
* Conversion of surgery from laparoscopy to open surgery.

Ages: 18 Years to 64 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 123 (Actual)
Dates: Start 2019-01-22 (Actual); Primary Completion 2021-03-20 (Actual); Study Completion 2021-04-30 (Actual)

PRIMARY OUTCOMES:
Pain Visual Analog Scale | It is measured preoperatively and after the end of the operation at the 30th minute, 12th hour and 24th hour (up to 24 hours). Change from baseline Pain Visual Analog Scale scores at 24 hours.
  The Visual Pain Scale is a scale of ten centimeters, created to inquire about the pain status of individuals. Zero indicates no pain while ten indicates the most severe pain. This chart is prepared as a blank line for self-evaluation and the prepared chart is read on the ruler.
Thermal Comfort Visual Analog Scale | It is measured before surgery and every half hour after surgery (up to 2 hours). The change in thermal comfort score before and within the first two hours after surgery is recorded.
  Horn et al. It is a visual assessment scale developed by. Thermal comfort is evaluated using a 100 mm long visual benchmark scale. Zero points represent the worst unbearable cold, 50 mm thermal comfort, 100 mm unbearable temperature. Objective responses of the patients were determined by making an evaluation from 0 to 100mm.
Body Temperature Scale | It is measured before surgery and every fifteen minutes after surgery (up to 2 hours). The change in Body Temperature Scale score before and within the first two hours after surgery is recorded.
  It is the measurement chart prepared by the researcher. Includes measurement of body temperature over time.

SECONDARY OUTCOMES:
Tremor Rating Scale | It is measured before and every 15 minutes after surgery (up to 1 hour). Changes in tremor from the first minute to an hour after surgery.
  Badjatia et al. it is a visual assessment scale developed by. The tremor intensity rating scale is a visual evaluation scale that is observed and evaluated by researchers. When the quality of the tremor is evaluated numerically; 0: no flickering; 1: tremor localized in the abdomen and neck; 2: tremors, including upper limbs; and 3: whole body tremors.
Hemoglobin Parameters Scale | The hemoglobin level is measured before surgery and at 24th hours after surgery (up to 24 hours). Change from baseline hemoglobin level scores at 24 hours.
  Hemoglobin Parameters include leves at blood. Indicates the intraoperative bleeding level.
International Normalized Ratio Parameters Scale | The Pt INR level is measured before surgery and at 1th hours after surgery (up to 1 hours). Change from preoperative Pt INR level at postoperative 1st hour.
  International Normalized Ratio Parameters include Pt INR leves at blood. Indicates the intraoperative bleeding risk of patients.

CONTACTS AND LOCATIONS:
Locations (1):
- Yozgat Bozok University Health Sciences Faculty, Yozgat, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No